CLINICAL TRIAL: NCT05252299
Title: Feasibility and Acceptability of Rolling Refresher Training for Caregivers on Proper Infant Car Seat Use, Version 4.0, July 12, 2018
Brief Title: Infant Car Seat Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, James Chamberlain, Emergency Medicine Physician, Children's National Research Institute
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 00013738
Record Dates: First submitted 2021-12-02; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Pediatric Car Seat Safety Training
Keywords: car seat; Pediatric; safety

STUDY DESIGN:
Intervention Model Description: Statistical power is not the goal for this pilot study; rather, we wish to obtain estimates of feasibility as a basis for a future randomized controlled trial. As such, we plan to enroll 30 caregivers in each group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Refresher Training Group (Experimental): This study will use telemedicine to facilitate an innovative use of "rolling refresher" training (RRT), a technique used in medical education to provide hands-on interactive training at regular intervals with the goal of improving psychomotor skills required for high stakes procedures such as cardiopulmonary resuscitation. This study seeks to interrogate our hypothesis that providing instruction on CSS use to caretakers via telemedicine every 3 months during the first year of an infant's life is feasible and acceptable to caregivers.
  Interventions: Other: Rolling Fresher Group
- Traditional Group (No Intervention): They leave the hospital without the additional training and under hospital's normal discharge plan

INTERVENTIONS:
Other: Rolling Fresher Group — The use of telemedicine to provide remote CSS installation instruction via audio and visual input by a Certified child passenger safety technician (CPST)
  Arms: Refresher Training Group

SUMMARY:
Motor vehicle crashes (MVCs) kill more children and young adults than any other single cause in the United States. Proper use of the child safety seat (car seat, or CSS) reduces the risk of death by 71% in infants, and to toddlers by 54%. While the rate of CSS use has increased across all age groups over the last few decades,91% of observed CSSs demonstrate serious installation errors in the newborn population and 62% in all ages.In addition, non-white children have higher rates of misuse and non-use of CSS compared to white children, and the proportion of unrestrained deaths from MVCs in black and Hispanic children is almost twice that of white children (45% vs 26%). Certified child passenger safety technicians (CPST) provide interactive training to families on how to install and correct errors in their child's CSS. The use of CPSTs through "car seat checks" has been successful in increasing participants' (caregivers) skills, knowledge, and confidence, and reducing errors in CSS use.

DETAILED DESCRIPTION:
Motor vehicle crashes (MVCs) kill more children and young adults than any other single cause in the United States. Proper use of the child safety seat (car seat, or CSS) reduces the risk of death by 71% in infants, and to toddlers by 54%. While the rate of CSS use has increased across all age groups over the last few decades,91% of observed CSSs demonstrate serious installation errors in the newborn population and 62% in all ages.In addition, non-white children have higher rates of misuse and non-use of CSS compared to white children, and the proportion of unrestrained deaths from MVCs in black and Hispanic children is almost twice that of white children (45% vs 26%). Certified child passenger safety technicians (CPST) provide interactive training to families on how to install and correct errors in their child's CSS. The use of CPSTs through "car seat checks" has been successful in increasing caregivers' skills, knowledge, and confidence, and reducing errors in CSS use. However, car seat checks are disproportionately accessed by parents who are white, middle or upper class, and college-educated and thereby are not serving as an effective solution for the racial disparities in CSS misuse. In addition, there are challenges: A one-time interaction with a CPST does not lead to sustained success in correction of CSS errors, with 40% of families demonstrating serious errors in CSS use just 4 months after training; and with only about 33,000 CPSTs nationally for over 40 million CSS-eligible children, the resources required for in-person CPSTs to be easily accessible to all families with CSS eligible children make broad dissemination difficult. Remote quarterly CSS instruction via telemedicine can perhaps alleviate these problems and make CPSTs more easily accessible to all, including low-income and non-white families. Preliminary research reveals that the use of telemedicine to provide remote CSS installation instruction via audio and visual input by a CPST is better than using the written instruction manual alone, and leads to increased parental self-efficacy. In addition, telemedicine has been successfully used to address racial disparities in the treatment of heart failure, acute stroke, and other disease processes.

This study will use telemedicine to facilitate an innovative use of "rolling refresher" training (RRT), a technique used in medical education to provide hands-on interactive training at regular intervals with the goal of improving psychomotor skills required for high stakes procedures such as cardiopulmonary resuscitation. This study seeks to interrogate the investigator's hypothesis that providing instruction on CSS use to participants via telemedicine every 3 months during the first year of an infant's life is feasible and acceptable to participants. The investigators plan to do this through three specific aims: (1) Identify perceived barriers and motivators of participants to receipt of instruction on proper CSS use, and tailor intervention details based on their input; (2) Measure the feasibility and acceptability of providing participant-centered RRT on CSS use in a diverse population, including non-white populations at risk for disparities; and (3) Measure the preliminary effectiveness of RRT on serious errors in CSS use, and the disparities in error rates. Results will be used to develop a randomized controlled trial to evaluate the impact of using telemedicine to provide RRT on CSS use and impact on the known racial disparities in CSS use.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking parents and/or caregivers of full-term newborns born at the George Washington University (GWU) Hospital, and
* Mother/child are discharged from GWU Hospital together
* Have regular access to a car, and
* Have access to a smartphone or tablet

Exclusion Criteria:

* Parents/caregivers who do not speak English or Spanish
* Mother and newborn are not discharged together
* Infant is premature (< 35 weeks gestational age) Parents/caregivers do not have access to smartphone or tablet
* Parents/caregivers do not have regular access to a car

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability of the car seat enhanced usual care and the intervention group | 1 year
  Both the enhanced usual care and the intervention groups will be provided an initial in-person car seat check prior to discharge from the nursery, which will include documentation and correction of errors and survey completion by participants. Rates of the feasibility outcomes (with 95% confidence intervals (CI's)) will be calculated. This is also measured by the retention of the participants in the year-long intervention.
The proportion of caregivers who made critical CSS use errors during CSS | 1 year
  Errors will be assessed as a dichotomous variable indicating whether or not any errors were made at each visit using repeated measures log-binomial regression. An interaction term between randomization group and time will be included in the model to estimate differences in slope (i.e. change in proportion of caregivers making errors) between the intervention and control groups over the course of the study. To explore differential effects by race/ethnicity, a three-way interaction term of group x race x time will be used to evaluate whether differences in slope between intervention and control groups differ by race/ethnicity (i.e. whether effects of the intervention are stronger in the non-white population).
The reduction in total number of CSS use errors | 1 year
  The CSS check will be provided by telemedicine for both the enhanced usual care and intervention groups at 0 and 9 months of age. The CSS check will be provided to the intervention group using telemedicine technology (Help Lightning) at 3, 6, and 9 months of age. Participants in both groups will have CSS use errors recorded with each interaction with a CPST. The intervention group will have errors recorded every 3 months, and the enhanced usual care group will have errors recorded at the 0 and 9 month car seat checks. Proportion of caregivers with critical errors, and total number of errors will be evaluated and compared between the intervention and control groups at the newborn, 12, 18 and, and 24 month points.

CONTACTS AND LOCATIONS:
Overall Officials: James Chamberlain, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- George Washington Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No